CLINICAL TRIAL: NCT04840849
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Nirsevimab in Healthy Chinese Adults
Brief Title: Evaluate the Pharmacokinetics, Safety, and Tolerability of Nirsevimab in Healthy Chinese Adults
Acronym: PK/ADA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: IQVIA RDS (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: D5290C00007
Record Dates: First submitted 2021-04-08; First posted 2021-04-12 (Actual); Results first posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2022-12

CONDITIONS: Evaluate PK Profile
Keywords: PK; safety; tolerability; Nirsevimab; healthy Chinese Adults; Respiratory Syncytial Viral (RSV)
MeSH Terms: interventions — nirsevimab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nirsevimab (Experimental): Nirsevimab single dose IM injection
  Interventions: Biological: nirsevimab
- Placebo (Placebo Comparator): Placebo single dose IM injection
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: nirsevimab — Drug: injection, a single fixed IM dose on day 1 only.
  Other Names: MEDI8897
  Arms: Nirsevimab
Other: Placebo — Placebo: injection, 0.9% (w/v) saline, a single fixed IM dose on day 1 only.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the Pharmacokinetics, Safety, Tolerability of Nirsevimab in Healthy Chinese Adults.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind, placebo-controlled study to evaluate the PK, safety and tolerability, and ADA of nirsevimab when administered as a single fixed IM dosage to healthy Chinese adult subjects. Enrolment is planned at a single study center in China. Approximately 24 subjects will be randomly assigned in a 3:1 ratio to receive nirsevimab (n = 18) or placebo (n = 6). All subjects will be followed for approximately 150 days after dosing to assess safety, PK, and ADA response.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 45 years
2. Weight ≥ 45 kg and ≤ 110 kg and Body Mass Index of 19 to 26 kg/m2
3. Healthy Chinese subjects (both male and female)
4. Normotensive
5. Normal electrocardiogram (ECG) within 28 days prior to Day 1

Exclusion Criteria:

1. Acute illness at study entry (pre-dose on Day 1)
2. Fever ≥99.5°F (37.5°C) on day of dosing
3. Any drug therapy within 14 days prior to Day 1 (except contraceptives).
4. Receipt of immunoglobulin or blood products within 6 months prior to study entry.
5. Receipt of any investigational drug therapy within 120 days prior to investigational product dosing or planned to receive any investigational drug therapy within 150 days after investigational product dosing.
6. Previous receipt of any marketed or investigational mAb.
7. Previous vaccination against RSV.
8. History of immunodeficiency or receipt of immunosuppressive medications during the prior year.
9. History of asthma.
10. History of autoimmune disorder.
11. Evidence of any systemic disease on physical examination.
12. Evidence of infection with hepatitis A, B, or C virus, syphilis, or human immunodeficiency virus.
13. Any clinically significant abnormal laboratory assessments at screening.
14. Pregnant or nursing mother.
15. Alcohol or drug abuse

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-11-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSP_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5290C00007&attachmentIdentifier=b6aa3e08-3421-4b30-801f-a40f95d79abb&fileName=CSP_Redacted.pdf&versionIdentifier=
- See also: SAP_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5290C00007&attachmentIdentifier=f6d7f5bc-9be5-4d1c-856c-dbcd3c6dfccc&fileName=SAP_Redacted.pdf&versionIdentifier=
- See also: CSR_Synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5290C00007&attachmentIdentifier=db59724f-6272-479b-84e4-14a1ec7327cb&fileName=CSR_Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase 1, placebo-controlled, study to evaluate pharmacokinetics (PK), safety, and tolerability of nirsevimab compared to placebo in healthy participants conducted at a single center in China.
Pre-assignment Details: This study consisted of a screening period (28 days) and treatment period (151 days). A total of 24 participants were randomized in a 3:1 ratio to receive either nirsevimab or placebo.
Groups:
- Nirsevimab: Participants received single fixed intramuscular (IM) dose of nirsevimab on Day 1.
- Placebo: Participants received single fixed IM dose of placebo matching with nirsevimab on Day 1.
Period: Overall Study
Arm/Group | Nirsevimab | Placebo
Started | 18 | 6
Completed | 18 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: As-treated population included all participants who were randomized into the study and received any amount of study treatment.
Groups:
- Nirsevimab: Participants received single fixed IM dose of nirsevimab on Day 1.
- Total: Total of all reporting groups
Arm/Group | Nirsevimab | Placebo | Total
Number analyzed (Participants) | 18 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (5.55) | 29.8 (4.71) | 29.3 (5.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 15 | 2 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 6 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 18 | 6 | 24

OUTCOME MEASURES:

1. Primary Outcome: Serum Concentrations of Nirsevimab
Description: Serum samples were collected at indicated timepoints to determine the serum concentration of nirsevimab.
Time Frame: Pre-dose on Day 1 and on Days 2, 4, 6, 8, 15, 31, 91, 151 post-dose.
Population: The PK population included all participants who received any dose of study treatment and had at least one measurable post-dose serum PK observation and for whom PK blood samples were assumed not to be affected by factors such as important protocol deviations (if any, determined prior to unblinding).
  Only participants who received nirsevimab were analyzed for PK outcome measures.
Measure: Mean (Standard Deviation); unit: micrograms/milliliter (mcg/mL)
Arm/Group | Nirsevimab
Number analyzed (Participants) | 18
micrograms/milliliter (mcg/mL)
  Pre-dose Day 1 | NA (NA) — NA indicates mean and standard deviation below the lower limit of quantitation of 0.5 mcg/mL
  Day 2 | 27.644 (5.819)
  Day 4 | 41.794 (8.447)
  Day 6 | 43.811 (8.291)
  Day 8 | 46.050 (12.484)
  Day 15 | 43.739 (7.236)
  Day 31 | 40.300 (5.391)
  Day 91 | 25.200 (3.694)
  Day 151 | 17.597 (3.854)

2. Primary Outcome: Maximum Observed Serum Concentration (Cmax) for Nirsevimab
Description: Cmax for nirsevimab was directly calculated from the individual concentration-time curve.
Time Frame: Pre-dose on Day 1 and on Days 2, 4, 6, 8, 15, 31, 91, 151 post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Nirsevimab
Number analyzed (Participants) | 18
mcg/mL | 46.882 (21.7)

3. Primary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) for Nirsevimab
Description: Tmax for nirsevimab was directly calculated from the individual concentration-time curve.
Time Frame: Pre-dose on Day 1 and on Days 2, 4, 6, 8, 15, 31, 91, 151 post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Nirsevimab
Number analyzed (Participants) | 18
days | 6.99 [4.91 to 29.90]

4. Primary Outcome: Area Under the Serum Concentration-Time Curve From Time 0 to 150 Days (AUC0-150) for Nirsevimab
Description: Area Under the Serum Concentration-Time Curve From Time 0 to 150 Days (AUC0-150) for Nirsevimab was calculated by linear up/log down trapezoidal summation.
Time Frame: Pre-dose on Day 1 and on Days 2, 4, 6, 8, 15, 31, 91, 151 post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*day/mL
Arm/Group | Nirsevimab
Number analyzed (Participants) | 18
mcg*day/mL | 4210.56 (13.6)

5. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibody (ADA) of Nirsevimab
Description: ADA positive was defined as any participant with a positive ADA result available at any time, including baseline and all post-baseline measurements; otherwise ADA negative.
Time Frame: Baseline (Day 1) and Days 31, 91 and 151
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Nirsevimab
Number analyzed (Participants) | 18
Participants
  Baseline (Day 1) | 0
  Day 31 | 0
  Day 91 | 0
  Day 151 | 0

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were collected from first date of study treatment administration (Day 1) up to 151 days.
Description: Treatment emergent adverse events were reported for As-treated population which included all participants who were randomized into the study and received any amount of study treatment.
Arm/Group | Nirsevimab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/6
Other Adverse Events (participants affected / at risk) | 5/18 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nirsevimab (N=18) | Placebo (N=6)
Haemoglobin decreased (Investigations) | 1 (1) | 1 (1)
Urobilinogen urine increased (Investigations) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Complement factor decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-12-04): https://cdn.clinicaltrials.gov/large-docs/49/NCT04840849/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT04840849/SAP_001.pdf